CLINICAL TRIAL: NCT01884129
Title: Prognostic Value of Circulating Tumor Cells in Patients With Locally Advanced and Metastatic/Recurrent Head and Neck Cancer
Brief Title: Prognostic Value of CTC in HNSCC Patients
Acronym: CTCHNSCC01
Status: Terminated | Type: Observational
Why Stopped: participants are no longer being examined or treated
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CTCHNSCC01; CMRPG3B0971~3 (Other Grant/Funding Number: CMRPG3B0971~3)
Record Dates: First submitted 2013-06-10; First posted 2013-06-21 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2013-02

CONDITIONS: Recurrence; Metastasis; Death
Keywords: Circulating tumor cells; Head and neck cancer; Squamous cell carcinoma; Survival; Prognosis
MeSH Terms: conditions — Recurrence; Neoplasm Metastasis; Death; Neoplastic Cells, Circulating; Head and Neck Neoplasms; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: None Retained — Blood samples were drawn by standard procedure, stored in EDTA-coating tubes in 4 degree temperature, then sent for CTCs counting and analysis.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
We hypothesized that the number of circulating tumor cells (CTCs) and molecular markers on CTCs could be a prognostic factor or predictive factor to patients with head neck cancer.

DETAILED DESCRIPTION:
1. Histologically or cytopathologically proven head and neck squamous cell carcinoma (HNSCC)
2. Disease status: locally advanced or recurrent/metastasized at initial presentation
3. Age >=20 years old
4. Could understand and signed the informed consents of this study
5. Enrolled patients were classified into three distinct subgroups:

   1. Patients underwent curative surgery followed by adjuvant chemoradiotherapy (CRT) because of some pathologic features such as positive margin, pathologic N2, and extracapsular spread (ECS) of involved lymph nodes indicating early relapse according to recommendation from National Comprehensive Cancer Network(NCCN) guidelines;
   2. Patients with advanced disease directly underwent definitive concurrent chemoradiotherapy(CCRT);
   3. Patients were to have palliative chemotherapy for existence of distant metastasis or poor general condition for definitive CCRT.
6. Blood samples were collected within 7 days before the first dose of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytopathologically proven head and neck squamous cell carcinoma Age ≥ 20 years. Measurable or evaluable disease according to Response Evaluation Criteria In Solid Tumors(RECIST) criteria.

Ability to sign informed consent.

Exclusion Criteria:

* Prior cancers within 5 years, except for non-melanoma skin cancers, and in situ cervical cancers.

Inability to comply with study and/or follow-up procedures.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Locally advanced or recurrent/metastatic head and neck cancer
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2012-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | one year
  Measure response or progression events via all available imaging studies, including Chest-Xray, CT scans, or MRI, PET study. The relationship between CTCs number and time from CTCs checkpoint to disease progression will be analyzed.

OTHER OUTCOMES:
Overall survival | one year
  All causes of death would be documented and the relationship between CTCs number and time from CTCs checkpoint to death will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hsun C Hsieh, M.D, M.S., Principal Investigator — Division of Hematology-Oncology, Department of Internal Medicine, Chang Gung Memorial Hospital at Linkou
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Hsieh JC, Lin HC, Huang CY, Hsu HL, Wu TM, Lee CL, Chen MC, Wang HM, Tseng CP. Prognostic value of circulating tumor cells with podoplanin expression in patients with locally advanced or metastatic head and neck squamous cell carcinoma. Head Neck. 2015 Oct;37(10):1448-55. doi: 10.1002/hed.23779. Epub 2014 Jul 24. PMID 24844673